CLINICAL TRIAL: NCT05744973
Title: Multi-level Predictors of Structural Racism and Discrimination and Associations With Health and Well-being Across the Life Course in Diverse Families
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: SRD
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Racially/Ethnically Diverse Families From Urban Settings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Minoritized populations face mutually reinforcing levels of structural disadvantage that contribute to poor health. Despite recognition that social and economic stratification, environmental conditions, and policy are critical determinants of health disparities, there has been limited effort in expanding interventions beyond the individual level to disrupt systemic causes of health. This is in part due to the challenges of describing how racism and discrimination have become systematized over time and across place.68 Studies that do examine SRD and health and well-being, focus on one level of SRD at a time, rather than examining multiple levels simultaneously. Also, the measurement of SRD at all levels has not been very detailed and more research is needed on the nuances of these experiences (e.g., frequency, timeframe, intensity). Finally, there is a need for more prospective longitudinal studies, as most research to date has been cross-sectional. In addition to comprehensively examining the four SRD levels, the current study will examine these multi- level predictors of SRD simultaneously, longitudinally, and across two sites to identify targets for multi-level interventions that will be more likely to be effective and sustainable.

ELIGIBILITY:
Inclusion Criteria:

* willingness to provide informed consent (parent/guardian), parental consent (parent/guardian) and assent (minor participants) and the ability for participants to comply with study requirements
* They are the child's primary caregiver, i.e., they are the adult who spends the largest proportion of time caring for the child (e.g., cleaning, feeding, etc.) or they spent an exactly equal proportion to another caregiver (e.g., parents each with 50% of childcare responsibilities).
* They reside in Athens-Clarke County or surrounding counties (i.e., Barrow, Jackson, Madison, Oglethorpe, and Oconee) served by the Piedmont Healthcare Coalition region
* Have access to a smartphone or other internet-connected device (e.g., iPad; home computer; laptop)
* Are able to read either English or Spanish

UMN site:

* participation in the original Family Matters Ecological Momentary Assessment sub-study
* did not withdraw from the Family Matters study
* ability to participate in an in-person visit (e.g., within driving distance to make an in-person visit)
* The original Family Matters study enrolled vulnerable populations including children, pregnant women, disadvantaged persons, and non-English speakers.

UGA site:

* Child has a racial/ethnic identity reported by the parent as Black, Hispanic, or White Reside in Athens-Clarke County or surrounding counties (i.e., Barrow, Jackson, Madison, Oglethorpe, and Oconee) served by the Piedmont Healthcare Coalition region
* Have access to a smartphone or other internet-connected device (e.g., iPad; home computer; laptop)
* Are able to read either English or Spanish
* Aged 8 to 18 years old

Exclusion Criteria:

* Medically necessary dietary restrictions (e.g., feeding tubes)
* BMI < 5%ile
* A diagnosis of a serious and persistent mental illness
* The child's parent/caregiver believes that the child is not developmentally able to participate in study components (e.g., severe autism)
* The family already has one parent or one child enrolled in the study
* There are no more availabilities in the family's census tract (limited to 10 households per tract). UGA also is interested in recruiting families from a range of census tracts in the Athens, GA area. If UGA finds that many families are coming from a few census tracts, they may restrict enrollment of new participants who are from those already-represented census tracts.

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: UMN:
  The study will be enrolling vulnerable populations, just as it did during the original study. To accommodate for this, children will be assented into the study and all participant materials will be translated into Spanish, Hmong, and Somali. Bilingual staff will be employed and able to assist participants whose reading skills are limited. The study will provide free parking to participants and compensate all participants (both parents and children) for their time spent on study processes.
  The study will enroll participants who happen to be pregnant and will not seek out pregnant adolescents. UGA: The University of Georgia site will follow the same process to accommodate vulnerable populations.
Sampling Method: Non-Probability Sample
Enrollment: 631 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
changes in cardiometabolic risk score | baseline to 18 months
  comprised of 5 cardiometabolic indicators of lower health - overweight status, triglyceride to HDL ratio, c-reactive protein , stage 1 or 2 hypertension, and elevated HbA1c >= 5.7across two time points 18 months apart collected in children and adults

SECONDARY OUTCOMES:
Change in Mental health (parent and child) | baseline to 18 months
  Change in depression scores using Kessler 6
Dietary intake | baseline to 18 months
  Change in modified HEI score
Physical Activity | baseline to 18 months
  Change in Sedentary Activity and Moderate/Vigorous Physical Activity using Godin Shephard

CONTACTS AND LOCATIONS:
Overall Officials: Jerica Berge, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Georgia, Athens, Georgia
  - University of Minnesota, Minneapolis, Minnesota